CLINICAL TRIAL: NCT07385326
Title: Effect of Umbilical Cord Clamping Method on Peripheral Blood Stem Cell Counts in Preterm Newborns: A Randomized Controlled Trial
Brief Title: Umbilical Cord Clamping Methods and Stem Cell Counts in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Era Tufan Benli (Other)
Responsible Party: Sponsor-Investigator, Era Tufan Benli, Principal Investigator, Dr. Sami Ulus Children's Hospital
Organization: Dr. Sami Ulus Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SUCCH-UCC-2015
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth; Umbilical Cord Clamping
Keywords: Preterm newborn; Umbilical cord clamping; Hematopoietic stem cells; Peripheral blood; Randomized study
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to three parallel groups based on umbilical cord management method.
Masking Description: Outcome assessors were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Cord Clamping (ICC) (Experimental): Umbilical cord clamped within 30 seconds after birth.
  Interventions: Procedure: Immediate Cord Clamping
- Delayed Cord Clamping (DCC) (Experimental): Umbilical cord clamped 60 seconds after birth.
  Interventions: Procedure: Delayed Cord Clamping
- Umbilical Cord Milking (UCM) (Experimental): Umbilical cord milked toward the infant before clamping.
  Interventions: Procedure: Umbilical Cord Milking

INTERVENTIONS:
Procedure: Immediate Cord Clamping — Clamping of the umbilical cord within 30 seconds after delivery.
  Arms: Immediate Cord Clamping (ICC)
Procedure: Delayed Cord Clamping — Clamping of the umbilical cord 60 seconds after delivery.
  Arms: Delayed Cord Clamping (DCC)
Procedure: Umbilical Cord Milking — Milking of a 20 cm segment of the umbilical cord toward the infant before clamping.
  Arms: Umbilical Cord Milking (UCM)

SUMMARY:
This study evaluates the effect of different umbilical cord clamping methods on peripheral blood hematopoietic stem cell counts in preterm newborns.

Preterm infants were randomly assigned to different umbilical cord clamping strategies as part of routine obstetric care. Peripheral blood samples were collected after birth to assess stem cell concentrations.

The aim of the study was to determine whether physiological cord management strategies could influence early hematologic adaptation in preterm infants. The study was conducted using standard clinical procedures without additional intervention beyond routine care.

DETAILED DESCRIPTION:
This prospective randomized study was conducted to investigate the impact of different umbilical cord clamping methods on peripheral blood hematopoietic stem cell counts in preterm newborns.

Eligible preterm infants were randomly allocated to one of the predefined umbilical cord clamping strategies according to the study protocol. All procedures were performed as part of standard obstetric and neonatal care, and no experimental intervention outside routine clinical practice was applied.

Peripheral blood samples were obtained following delivery, and hematopoietic stem cell concentrations were analyzed using standard laboratory methods. The primary outcome was the comparison of stem cell counts between the different cord clamping groups.

The study was initiated and completed in 2015, prior to mandatory prospective clinical trial registration requirements. Ethical approval was obtained from the relevant institutional ethics committee, and informed consent was obtained from parents or legal guardians before participation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates born between 28+0 and 36+6 weeks of gestation.
* Infants born at a single tertiary referral center.
* Written informed consent obtained from parents prior to delivery.

Exclusion Criteria:

* Major fetal congenital anomalies.
* Perinatal asphyxia.
* Requirement for advanced neonatal resuscitation at birth.
* Undetermined gestational age.
* Gestational age less than 28 weeks.

Min Age: 0 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neonatal Hemoglobin Level | Within first 24 hours after birth
  Comparison of neonatal hemoglobin levels among immediate cord clamping, delayed cord clamping, and umbilical cord milking groups.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Ceyhan, Dr., Principal Investigator — Department of Gynecology and Obstetrics, Lokman Hekim University, Faculty of Medicine,
Locations (1):
- Department of Gynecology and Obstetrics, Lokman Hekim University, Faculty of Medicine,, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No